CLINICAL TRIAL: NCT02337777
Title: The Study of Functional Magnetic Resonance Imaging in Abdominal and Pelvic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Hu Daoyu, PhD,Professor, Tongji Hospital
Other Study IDs: S097
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pelvic Diseases; Abdominal Diseases
Keywords: Magnetic Resonance Imaging; Magnetic Resonance Angiography; Diffusion Tensor Imaging; IDEAL; T2* mapping; Magnetic ResonanceCine; BOLD; phase contrast; diffusion-weighted imaging; Functional Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to study the diagnostic efficiency of functional magnetic resonance imaging in Abdominal and Pelvic Diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients with abdominal or pelvic diseases who provide informed consent
* Healthy Volunteers

Exclusion Criteria:

* claustrophobic
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with abdominal or pelvic diseases who provide informed consent Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 10years

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical college of Huazhong Universitity of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Tang H, Wang Z, Wang L, Hu X, Wang Q, Li Z, Li J, Meng X, Wang Y, Hu D. Depiction of transplant renal vascular anatomy and complications: unenhanced MR angiography by using spatial labeling with multiple inversion pulses. Radiology. 2014 Jun;271(3):879-87. doi: 10.1148/radiol.14131800. Epub 2014 Mar 3. PMID 24592960
- [Result] Wang YC, Hu DY, Hu XM, Shen YQ, Meng XY, Tang H, Li Z. Assessing the Early Response of Advanced Cervical Cancer to Neoadjuvant Chemotherapy Using Intravoxel Incoherent Motion Diffusion-weighted Magnetic Resonance Imaging: A Pilot Study. Chin Med J (Engl). 2016 Mar 20;129(6):665-71. doi: 10.4103/0366-6999.177995. PMID 26960369
- [Result] Wang Y, Li Z, Meng X, Hu X, Shen Y, Morelli J, Lin H, Zhang Z, Hu D. Nonmuscle-invasive and Muscle-invasive Urinary Bladder Cancer: Image Quality and Clinical Value of Reduced Field-of-view Versus Conventional Single-shot Echo-planar Imaging DWI. Medicine (Baltimore). 2016 Mar;95(10):e2951. doi: 10.1097/MD.0000000000002951. PMID 26962794